CLINICAL TRIAL: NCT06154473
Title: Assessment of Patients Undergoing Cardiac Surgery and Admitted to the Intensive Care Unit: an Observational, Prospective, Multicenter Study
Brief Title: Assessment of Patients Undergoing Cardiac Surgery and Admitted to the Intensive Care Unit
Acronym: BraSIS-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: 5350-22
Record Dates: First submitted 2023-07-25; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Disease; Cardiac Ischemia; Cardiac Valve Disease
Keywords: cardiac surgery; anesthesia; critical care; mortality; epidemiology
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open heart surgery: Cohort of patient undergoing an open heart surgery. Open heart surgery is defined as a surgical procedure that involves making an incision in the chest to opening the chest wall to access and operate on the heart. The study will include patients who undergo valve repair, valve replacement, or coronary artery bypass grafting. In addition, combined surgery, define as valve surgery in combination with coronary artery bypass grafting, will also be included. Heart transplant will not be included.
  Interventions: Procedure: Open heart surgery group.
- Percutaneous cardiovascular surgery: Cohort of patient undergoing a percutaneous cardiovascular surgery. Percutaneous cardiovascular surgery is defined as a surgical procedure that involves making an incision in the skin to use a catheter-based approach to access and operate on the heart. The study will include patients who undergo transcatheter aortic valve implantation, valve in valve transcatheter aortic valve implantation and transcatheter mitral-valve repair or replacement.
  Interventions: Procedure: Percutaneous cardiovascular surgery group.

INTERVENTIONS:
Procedure: Open heart surgery group. — Patients undergoing open heart surgery.
  Groups: Open heart surgery
Procedure: Percutaneous cardiovascular surgery group. — Patients undergoing percutaneous cardiovascular surgery.
  Groups: Percutaneous cardiovascular surgery

SUMMARY:
The objective of this study is to investigate the incidence of death and early postoperative complications, identify potential risk factors, and examine the demographic characteristics of patients and epidemiology of cardiovascular procedures. Our hypothesis is that gaining a more comprehensive understanding of the characteristics of patients who undergo cardiac surgery has the potential to improve outcomes for this patient profile. Thus, information was sought regarding the patient characteristics, surgeries performed, anesthesia administered, incidence of intraoperative and postoperative complications, and risk factors associated with complication and mortality in the ICU. The main questions it aims to answer are:

* Incidence of mortality or severe postoperative complications that occur within the first 3 postoperative days or until discharge from the ICU.
* Risk factors associated with severe complications in patients who undergo cardiac surgery.
* Characteristics of patients, anesthesia and surgical procedures performed
* Incidence of severe intraoperative complications and moderate postoperative complications
* Evaluate the influence of accumulated fluid balance on outcomes, mortality, and length of ICU stay.
* Evaluate mortality in the ICU.
* Describe the risk factors associated with mortality.

DETAILED DESCRIPTION:
BACKGROUND The results of procedures in patients undergoing cardiovascular surgery are significantly influenced by preoperative risk factors and adequate perioperative management. Therefore, it is essential to develop tools and strategies that provide improvements in care to minimize complications.

SAMPLE SIZE CALCULATION The aim is to consecutively include 500 patients who undergo cardiac surgery. The incidence of death or severe postoperative complications in cardiovascular surgery during the first 3 postoperative days or until discharge from the ICU is approximately 20%. Therefore, with the inclusion of 500 patients, it will be possible to create a robust regression model by adding 10 independent variables.

PRIMARY OBJECTIVE Outcome composed of mortality or severe postoperative complications within the first 3 postoperative days or until ICU discharge, whichever occurs first. Severe postoperative complications are: stroke, septic shock, unscheduled urgent or emergency surgical reoperation, cardiovascular complications, hematological complications, pulmonary complications, and renal complications.

Cardiovascular complications: acute myocardial infarction, unplanned use of circulatory assist device, cardiac arrest with return of spontaneous circulation, severe hemodynamic instability.

Hematologic complication: severe bleeding. Pulmonary complications: acute respiratory distress syndrome (ARDS) with partial pressure of oxygen (PaO2) / inspired oxygen fraction (FiO2) ratio ≤ 250 (refractory to rescue maneuvers and ventilatory adjustment that persists for more than 1 hour), re-intubation in an unplanned manner.

Renal complications: Kidney Disease: Improving Global Outcomes (Kdigo) score ≥ 2 or renal replacement therapy.

Severe hemodynamic instability was defined as: use of norepinephrine ≥0.1 mcg/kg/min for more than 2 hours; or adrenaline ≥0.1 mcg/kg/min for more than 2 hours; or dose-independent combination of norepinephrine and adrenaline for more than 2 hours; or dose-independent combination of norepinephrine and vasopressin for more than 2 hours. It is important to note that there is no consensus on the definition of severe hemodynamic instability in the postoperative period of patients undergoing cardiac surgery. The definition of severe hemodynamic instability was made after literature review and extensive discussion with the executive committee of the BraSIS 2 trial.

Acute myocardial infarction is recommended diagnosis using the universal type 5 infarction classification: troponin elevation 10 times the 99th percentile.

Major bleeding is defined as a fall ≥ 2g/dl hemoglobin or transfusion of 2 red blood cells concentrates without an increase in hemoglobin value or bleeding associated with a fall in systolic blood pressure value ≥10 millimeter of mercury (mmHg) when the patient assumes the orthostatic position or a spontaneous fall in systolic blood pressure ≥ 20 mmHg or an increase in heart rate ≥ 20 beats per minute.

The diagnosis of ARDS was made by using the Berlin definition. To diagnose ARDS using the Berlin definition, the respiratory failure could not fully be explained by cardiac failure or volume overload. To exclude volume overload secondary to cardiac failure, it is suggested to use B-type natriuretic peptide (BNP) or N-terminal pro B-type natriuretic peptide (NT-proBNP) in combination with echocardiography to assess cardiac function.

STATISTICAL ANALYSIS Data will be collected as part of routine clinical care. Patient characteristics will be compared and described by appropriate methods. Histogram and Kolmogorov-Smirnov test will be used to evaluate the distribution pattern of continuous numerical variables. Qualitative variables will be expressed as proportions, quantitative variables will be expressed as mean ± standard deviation or as median and interquartile range when appropriate.

Continuous variables will be analyzed with Student's t-test, analysis of variance, Mann-Whitney U test, Kruskal-Wallis test, or Friedman test as appropriate. Categorical variables will be analyzed with chi-square test or Fisher's exact test as appropriate.

Analyses of time dependent variables will be evaluated using the paired t-test (or Wilcoxon signed rank test in case of non-normal distribution) if time effect is detected, Cox regression and visualized by Kaplan-Meier curve.

Comparisons between and within group will be performed using analysis of variance (ANOVA) and post-hoc analyses for continuous variables. The multiple logistic regression model will be used to identify independent risk factors for postoperative complications. Sub-groups of patients undergoing open heart surgery and patients undergoing percutaneous cardiovascular surgery will be analyzed separately.

The following subgroup analyses will be performed: patients with prior use of circulatory assist devices compared to patients without prior use of such devices, patients with prior use of vasoactive drugs compared to patients without preoperative use, comparison between types of cardioplegic solutions used, comparisons between types of circulatory assist devices, impact of CPB time on mortality and postoperative complications, impact of intraoperative use of etomidate. All significance probabilities (p-values) presented will be two-tailed. The p-values will be considered statistically significant when smaller than 0.05 or 95% confidence interval (CI) values that do not cross the number 1.0. Bonferroni correction will be used for multiple comparisons in post hoc tests. R version 4.0.0 software (R Foundation for Statistical Computing, Austria) and Python programming language (version 3.10, python.org) will be used to perform the analyses.

ADVERSE EVENTS The study does not present additional risks to those expected for patients undergoing cardiac surgery. The only anticipated risk would be a breach of data confidentiality, which will be mitigated as described in the data confidentiality item. Adverse events are defined as an unwanted experience suffered by a patient during the study, whether or not related to the proposed interventions. All adverse events must be reported to the research ethics committee that approved the trial. It is emphasized that mortality in a patient undergoing cardiac surgery is an event frequently encountered in this patient population, and although it is an unwanted event, it will not be defined as an adverse event. A severe adverse event is any unfavorable medical occurrence or effect that results in

* Life threatening (during the occurrence of the event).
* Requires hospitalization or prolongs the length of stay for patients already hospitalized.
* Significant or persistent physical disability.
* Any new event that affects patient safety, such as an unexpected outcome of the test drug, lack of efficacy of the test drug, or increased safety found in another drug similar to the study drug recently found in animal studies, etc.

REGULATORY STATUS The study will be conducted in accordance with the principles of the Declaration of Helsinki and in accordance with the Medical Research Involving Humans Act.

APPROVAL FROM ETHICS AND REGULATORY AUTHORITIES The study will be performed according to the national and international guidelines. The Institutional Review Board of the Hospital Israelita Albert Einstein has approved this study (CAAE: 69330823.1.0000.0071). The participating centers will not initiate the study until they have obtained approval from their respective local Institutional Review Boards.The need for informed consent is determined by the Institutional Review Board of each participating center.

CONFIDENTIALITY OF DATA The patient and the investigating center will be identified by the corresponding number on the electronic data collection form. Researchers will keep the data obtained from the medical record confidential and store it in cabinets with restricted access. The anonymity of all data in interim and final reports will be ensured. The data will be treated confidentially, and sites should keep all data stored for the length of the study and for as long as local regulations allow. After the designated time, data should be incinerated. Loss of data confidentiality is possible due to access to patient data. However, staff undertakes to take every care to ensure confidentiality of the data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years or older).
* Cardiac surgeries requiring postoperative care in the ICU.

Exclusion Criteria:

* Exclusive palliative care or advance directive expressing desire for limitation of life support (cardiopulmonary resuscitation, invasive mechanical ventilation, renal replacement therapy).
* Moribund patient.
* Surgery for implant of cardiac implantable electronic device (implantable cardioverter defibrillator, cardiac pacemaker).
* Patients previously included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Centers with experience in cardiac surgery will be invited to participate in the study. It is planned that patients undergoing cardiac surgery will be included consecutively during the study period, which will be determined later. The study population will consist of patients undergoing open heart surgery or percutaneous cardiovascular surgery, and the following surgeries will be included: valve repair (or replacement) and/or coronary artery bypass grafting.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Mortality or severe postoperative complications within the first 3 postoperative days or until ICU discharge, whichever occurs first | Within the first 3 postoperative days or until ICU discharge, whichever occurs first, assessed up to 3 postoperative days
  Severe postoperative complications are: stroke, septic shock, unscheduled urgent or emergency surgical reoperation, cardiovascular complications, hematological complications, pulmonary complications, and renal complications

SECONDARY OUTCOMES:
Evaluate the characteristics of the patients | Within the first 3 postoperative days or until ICU discharge, whichever occurs first, assessed up to 3 postoperative days
  Describe demographic characteristics of the patients
Describe the surgeries performed | Within the first 3 postoperative days or until ICU discharge, whichever occurs first, assessed up to 3 postoperative days
  Describe the type of surgeries performed. Description of the surgery as: emergency, urgent and elective surgery; open heart surgery or percutaneous cardiovascular surgery; valve repair (or replacement) and/or coronary artery bypass grafting
Describe the anesthesia performed | Within the first 3 postoperative days or until ICU discharge, whichever occurs first, assessed up to 3 postoperative days
  The following anesthesia modalities will be considered and collected: general anesthesia, combined general anesthesia (general anesthesia and neuroaxis block) and sedation
Evaluate the incidence of severe intraoperative complications | Within the first 3 postoperative days or until ICU discharge, whichever occurs first, assessed up to 3 postoperative days
  The following severe intraoperative complications will be considered and collected: bronchospasm or difficulty with respiratory support, failure to exit cardiopulmonary bypass (CPB), cardiac arrest with return of spontaneous circulation, and excessive blood transfusion (≥ 4 units of packed red blood cells)
Assess the incidence of other postoperative complications (not included in the primary endpoint) | Within the first 3 postoperative days or until ICU discharge, whichever occurs first, assessed up to 3 postoperative days
  The following postoperative complications will be considered and collect: cardiovascular; pulmonary; neurological, gastrointestinal and metabolic
Evaluate the influence of fluid balance on ICU mortality | Within the first 3 postoperative days or until ICU discharge, whichever occurs first, assessed up to 3 postoperative days
  Evaluate the influence of fluid balance on ICU mortality. Determine if the increase in fluid balance during the ICU stay is associated with the increase in ICU mortality.
Assess the length of stay in the ICU | Within the first 3 postoperative days or until ICU discharge, whichever occurs first, assessed up to 3 postoperative days
  Calculated from the date and time of admission and date and time of actual ICU discharge (discharge or death)
Evaluate the risk factors associated with ICU mortality | Within the first 3 postoperative days or until ICU discharge, whichever occurs first, assessed up to 3 postoperative days
  To construct a logistic regression model to identify risk factors associated with increased ICU mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Renato CF Chaves, MD, MBA., Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The study database will be accessible to other researchers as part of our plan. The database will be kept under the custody of the study coordinators, and its access could be allowed to third parties after evaluation of the proposal accompanied by a statistical analysis plan and execution of a Data Sharing Agreement. Once the agreement is in place, the database will be made available in an anonymized form. Should be emphasize that no data that allows future identification of the patient will be share. Example of data that will not be share: name, date of birth, individual registration number as Individual Taxpayer Registration (CPF), and medical record number. Each individual requesting access to the database must formally commit to notifying the executive committee of the study of any information that allows the identification of the patient in the database. For more information or to submit a request, please contact renato.carneiro@einstein.br
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting immediately after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal, review and approval of a statistical analysis plan and execution of a data sharing agreement. No data that allows future identification of the patient will be publicly available. For more information or to submit a request, please contact renato.carneiro@einstein.br

REFERENCES:
- [Derived] Vasconcelos NNB, Chaves RCF, Pellegrino CM, Souza GM, Queiroz VNF, Barbas CSV, Takaoka F, Cordioli RL, Mangini S, Papa FV, Guimaraes HP, Pereira AJ, Serpa Neto A, Gulinelli A, Legal AC, Jaoude CVG, Paolinelli E, Lineburger EB, Albuquerque ECF, Ferreira Filho EG, Hohmann FB, Galdino F, Vianna FSL, Dall'Orto FTC, Tramujas L, Silva LRP, Goncharov M, Gottardo PC, Rabello Filho R, Midega TD, Galindo VB, Quintao VC, Veiga VC, Correa TD, Silva Junior JM. Multicenter observational study of patients who underwent cardiac surgery and were hospitalized in an intensive care unit (BraSIS 2): study protocol and statistical analysis plan. Crit Care Sci. 2025 Mar 10;37:e20250222. doi: 10.62675/2965-2774.20250222. eCollection 2025. PMID 40072977